CLINICAL TRIAL: NCT01493362
Title: Imaging the Dopamine Systems in Bulimia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5175; R01MH079397 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2011-11

CONDITIONS: Eating Disorders
Keywords: Bulimia Nervosa; PET Imaging; Dopamine
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Participants with Bulimia Nervosa
- 2: Participants who are healthy controls

SUMMARY:
This study will use positron emission tomography imaging to investigate the dopamine systems in people with bulimia nervosa.

ELIGIBILITY:
Inclusion Criteria:

Participants with BN:

* Meets DSM-IV criteria for BN
* Sufficiently medically and psychiatrically stable to participate in research

Health Control Participants:

* No current or past psychiatric illness
* Between 80% and 120% of ideal body weight

Exclusion Criteria:

All participants:

* Current use of psychotropic medication such as anti psychotics or antidepressants
* Pregnant or breastfeeding
* history of substance abuse
* Significant medical illness
* High blood pressure (resting systolic blood pressure greater than 150mmHg and diastolic blood pressure greater that 90 mmHg)
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder as defined by DSM-IV
* Metal implants or paramagnetic objects contained within the body that may interfere with the MRI scan, as determined in consultation with a neuroradiologist and according to specified reference book guidelines
* Exposed to radiation in the workplace or has had a nuclear medicine procedure during the 1 year before study entry
* Previous adverse reaction to psycho stimulants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include people with bulimia nervosa seeking inpatient or outpatient treatment and people who will act as healthy control participants
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
D2 receptor density | Measured at baseline
DA release in the striatum | Measures after Mythlyphenidate challenge

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States